CLINICAL TRIAL: NCT06461026
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety, Tolerability, and Pharmacokinetics of L9LS in Infants in Mali and to Evaluate the Impact of L9LS on Subsequent R21/Matrix-MTM Vaccine Immunogenicity
Brief Title: L9LS MAb in Malian Infants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); University of Washington (Other); Harvard School of Public Health (HSPH) (Other); Indiana University School of Medicine, Indiana University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024/158/CE/USTTB
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 mg of L9LS (Experimental): Participants will receive a dose of 150 mg of L9LS.
  Interventions: Biological: L9LS
- Placebo (normal saline) (Placebo Comparator): Participants will receive placebo of Normal Saline for comparison.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: L9LS — Administered intramuscularly one time.
  Arms: 150 mg of L9LS
Other: Normal Saline — Administered intramuscularly one time.
  Arms: Placebo (normal saline)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of L9LS in infants in Mali and to evaluate the impact of L9LS on subsequent R21/Matrix-MTM vaccine immunogenicity.

DETAILED DESCRIPTION:
This is an age-stratified, randomized, double-blind, placebo-controlled trial evaluating the safety, tolerability, and pharmacokinetics (PK) of 1-time intramuscular (IM) administration of the monoclonal antibody (MAb) L9LS to healthy Malian infants aged 1 to 12 months, followed by an assessment of the impact of L9LS on the immunogenicity of subsequent administration of the R21/Matrix-MTM vaccine. The study hypotheses are that L9LS will be safe and will not impact the immunogenicity of the R21/Matrix-MTM vaccine. During the beginning of the 6-month malaria season (approximately August and September at the study site), 180 participants will be enrolled and randomized 1:1 to receive 150 mg of L9LS (n=90) or normal saline placebo (n=90). Randomization of participants in each arm will be age-stratified (1 to 4 months, n=60; >4 to 8 months, n=60; >8 to 12 months, n=60). The safety of L9LS will be assessed within each of the 3 age strata. Participants will be followed at study visits 1, 3, 7, 14, 21, and 28 days later, and once every 4 weeks thereafter through study day 280 (40 weeks). Approximately 5 months after receiving L9LS or placebo, all participants will receive the R21/Matrix-MTM vaccine as 3 total doses given 4 weeks apart as per World Health Organization (WHO) recommendations and the anticipated Malian vaccination guidelines. Primary study assessments include medical history, physical examination, and blood collection to assess antibody responses to the R21/Matrix-MTM vaccine, L9LS PK, anti-drug antibody (ADA) assessments, identification of Plasmodium falciparum (Pf) infection by microscopic examination of thick blood smears and reverse transcription polymerase chain reaction (RT-PCR), and other research laboratory evaluations. Through their local provider, all participants 3 months and older will be offered 4 rounds of seasonal malaria chemoprevention (SMC) as a monthly 3-day treatment course of sulfadoxine-pyrimethamine plus amodiaquine (SPAQ), as it is the standard of care in Mali for malaria prevention in children 3 months to 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥1 to ≤12 months at enrollment.
2. Born at ≥37 weeks gestation.
3. Parent and/or guardian able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history.
5. Parent and/or guardian able to provide informed consent.
6. Willing to have blood samples and data stored for future research.
7. Resides in or near Kalifabougou, Faladje, or Torodo, Mali, and available for the duration of the study.

Exclusion Criteria:

1. Body weight <3.5 kg.
2. Behavioral, cognitive, or psychiatric disease in the parent and/or guardian that in the opinion of the investigator affects the ability of the parent and/or guardian to understand and comply with the study protocol.
3. Any fever (≥ 37.5°C, regardless of route) or acute illness within 7 days prior to randomization.
4. Clinically significant congenital anomaly or documented or suspected serious medical illness (e.g., history of epilepsy), serious congenital anomaly, or immediate life-threatening condition in the infant that may interfere with the ability to complete study requirements, as judged by the examining clinician.
5. Prior history of a suspected or actual acute life-threatening event.
6. Receipt of any blood products, monoclonal or polyclonal antibody/immunoglobulin (for example, hepatitis B immune globulin, intravenous immunoglobulin) or anticipated use during the study.
7. Any acute or chronic illnesses known in the mother during her pregnancy.
8. Parental study comprehension examination score of <80% correct or per investigator discretion.
9. Hemoglobin, WBC, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Participants may be included at the investigator's discretion for "not clinically significant" values.)
10. ALT or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Participants may be included at the investigator's discretion for "not clinically significant" values.)
11. Mother and/or infant infected with HIV.
12. Sickle cell disease by testing. (Note: Known sickle cell trait is NOT exclusionary.)
13. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies.
14. Receipt of any investigational product within the past 30 days.
15. Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.)
16. History of a severe allergic reaction or anaphylaxis.
17. Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
18. Pre-existing autoimmune or antibody-mediated diseases including but not limited to systemic lupus erythematosus or autoimmune thrombocytopenia.
19. Known immunodeficiency syndrome.
20. Known asplenia or functional asplenia.
21. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
22. Previous receipt of the R21/Matrix-MTM vaccine.
23. Previous receipt of an investigational malaria vaccine or monoclonal antibody.
24. Clinical signs of malnutrition.
25. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of an individual participating in the trial, interfere with the evaluation of the study objectives, or render the participant unable to comply with the protocol.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of local and systemic AEs occurring within 7 days after the administration of study agent. | Measured through Day 7
Severity of local and systemic AEs occurring within 7 days after the administration of study agent. | Measured through Day 7
Measurement of study agent in sera of recipients. | Measured day 7, 28, 84, 140, 196 and 280

SECONDARY OUTCOMES:
Total IgG anti-NANP antibody titers measured by ELISA. | Measured 28 days and 84 days after the third R21/Matrix-MTM vaccination.
Measurement of Anti-Drug Antibodies (ADA) to L9LS in sera of recipients. | Measured at day 28, 224 and 280

CONTACTS AND LOCATIONS:
Overall Officials: Peter Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH); Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMOS)
Locations (3):
- Mali (3):
  - Faladje MRTC Clinic, Faladié, Koulikoro
  - Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro
  - Torodo MRTC Clinic, Torodo, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study for future research will be shared as follows:
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
  * De-identified results or data in publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: Data will be shared at the time of publication or shortly thereafter.
Access Criteria: Data from this study may be requested from other researchers indefinitely after the completion of the primary endpoint by contacting Laboratory of Immunogenetics.